CLINICAL TRIAL: NCT01811589
Title: Randomized Controlled Multi-center Trial Comparing the Ventricular Catheter Location Between Instrument Guided and Freehand Placement.
Brief Title: Guided Application of Ventricular Catheters
Acronym: GAVCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H1221
Record Dates: First submitted 2013-03-13; First posted 2013-03-14 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Hydrocephalus
Keywords: ventricular catheter, hydrocephalus, shunt, brain disease
MeSH Terms: conditions — Hydrocephalus; Brain Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thomale-Guide (Experimental): Positioning of ventricular catheter with the Thomale-Guide instrument
  Interventions: Device: Thomale-Guide
- Free-hand (Other): Ventricular catheter placement without a guidance (free-hand)
  Interventions: Other: Free-hand

INTERVENTIONS:
Device: Thomale-Guide — Ventricular catheter placement with the Thomale-Guide instrument
  Arms: Thomale-Guide
Other: Free-hand — Ventricular catheter placement without a guidance (free-hand)
  Arms: Free-hand

SUMMARY:
Failure of ventricular catheters remains a significant problem in patients with hydrocephalus. The purpose of this study is to determine whether the use of a simple instrument assisted by a smart phone application software can achieve a more precise placement of ventricular catheters than the standard free-hand placement technique.

DETAILED DESCRIPTION:
Free-hand placement of ventricular catheters (VC) is reported to be inaccurate in 10-40%. Furthermore, there is evidence that the quality of VC positioning is correlating with the risk for proximal shunt obstruction. Ultrasound or neuronavigation are used in order to improve to placement. However, they are associated with significant technical efforts and increased time.

In this study a simple instrument assisted by a smart phone application software is used in order to achieve precise placement of ventricular catheters. The results are compared with the standard free-hand procedure. Patients requiring a ventricular catheter are randomized to one of the two treatments. The primary outcome parameter is a qualitative and quantitative assessment of the position of the ventricular catheter on a post-operative image. The evaluation of the primary criteria is performed by a radiologist blinded to the randomization arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a permanent ventricular catheter for the treatment of CSF (cerebrospinal fluid) - circulation disorder or another disease (ventricular shunt oder Ommaya/Rickham-Reservoir)
* Frontal occipital horn ratio (FOHR) < 0.5
* Use of a new puncture channel
* Frontal access to the ventricles
* Patient´s informed consent

Exclusion Criteria:

* Known unevenness of the skull at the entry point
* Slit ventricles; Frontal and occipital horn width ratio (FOHWR) < 0.05
* Participation in another clinical trial with interfering endpoints

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Rate of he primary successful ventricular catheter placement with a Grade I or Grade I b and location in the ipsilateral ventricle | Within the first 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich W Thomale, PD Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (9):
- Germany (9):
  - Charité University Hospital, Division of Pediatric Neurosurgery, Berlin
  - Trauma Hospital Berlin, Clinic for Neurosurgery, Berlin
  - University Hospital Düsseldorf, Clinic for Neurosurgery, Düsseldorf
  - Univeristätsmedizin Göttingen, Neurochirurgie, Göttingen
  - Medizinische Hochschule Hannover, Neurochirurgie, Hanover
  - Heidelberg University Hospital, Department of Neurosurgery, Heidelberg
  - Klinikum Kassel GmbH / Department of Neurosurgery, Kassel
  - Dietrich-Bonhoeffer-Klinikum / Department of Neurosurgery, Neubrandenburg
  - University Hospital Tübingen, Department of Neurosurgery, Tübingen

REFERENCES:
- [Background] Thomale UW, Knitter T, Schaumann A, Ahmadi SA, Ziegler P, Schulz M, Miethke C. Smartphone-assisted guide for the placement of ventricular catheters. Childs Nerv Syst. 2013 Jan;29(1):131-9. doi: 10.1007/s00381-012-1943-1. Epub 2012 Oct 23. PMID 23089936
- [Result] Thomale UW, Schaumann A, Stockhammer F, Giese H, Schuster D, Kastner S, Ahmadi AS, Polemikos M, Bock HC, Golz L, Lemcke J, Hermann E, Schuhmann MU, Beez T, Fritsch M, Orakcioglu B, Vajkoczy P, Rohde V, Bohner G. GAVCA Study: Randomized, Multicenter Trial to Evaluate the Quality of Ventricular Catheter Placement with a Mobile Health Assisted Guidance Technique. Neurosurgery. 2018 Aug 1;83(2):252-262. doi: 10.1093/neuros/nyx420. PMID 28973670
- [Derived] Schaumann A, Thomale UW. Guided Application of Ventricular Catheters (GAVCA)--multicentre study to compare the ventricular catheter position after use of a catheter guide versus freehand application: study protocol for a randomised trail. Trials. 2013 Dec 12;14:428. doi: 10.1186/1745-6215-14-428. PMID 24330776